CLINICAL TRIAL: NCT06439706
Title: Assessing the Feasibility and Acceptability of Juntas Contra el Virus Del Papiloma Humano, an HPV Self-sampling Intervention for Underscreened Latinas
Brief Title: HPV Self-sampling for Underscreened Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Pennsylvania Breast Cancer Coalition (Unknown)
Responsible Party: Principal Investigator, Carolyn Fang, PhD, Associate Director of Population Science, Fox Chase Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 23-1027
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Uterine Cervical Neoplasm
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mailed Kit Only Control (Active Comparator): Participants receive an HPV self-sampling kit in the mail with instructions on how to self-collect a sample and return it to the lab for testing.
  Interventions: Behavioral: HPV Self-Sampling
- Education Plus Mailed Kit (Experimental): Participants receive information about cervical cancer risks and screening guidelines in a small-group format with a bilingual health educator. Participants also receive an HPV self-sampling kit in the mail with instructions on how to self-collect a sample and return it to the lab for testing.
  Interventions: Behavioral: HPV Self-Sampling; Behavioral: Group Education

INTERVENTIONS:
Behavioral: HPV Self-Sampling — HPV self-sampling kit
Behavioral: Group Education — Small-group education led by bilingual health educator
  Arms: Education Plus Mailed Kit

SUMMARY:
The goal of this study is to learn if women of Hispanic/Latina ethnicity are willing to self-collect a cervico-vaginal sample for HPV testing. The main question the study will answer is:

• Does a brief educational intervention increase the feasibility and acceptability of HPV self-sampling among Hispanic/Latina women?

The study team will compare whether including a brief educational intervention with a mailed HPV self-sampling kit is more acceptable than receiving a mailed HPV self-sampling kit alone.

Participants will be asked to complete surveys at study entry (baseline) and then randomized to receive only the HPV self-sampling kit, or the kit plus a small group education that meets with a bilingual health educator.

Participants will then be contacted about one-month later to complete a follow-up survey. The study team will also measure the number of participants in each group who self-collect a sample and mail it in for HPV testing.

DETAILED DESCRIPTION:
The study team will recruit a sample of underscreened Latinas (n=100) who will be randomly assigned to either the educational intervention (n=50) or a control condition (n=50). Feasibility will be measured through study enrollment and intervention completion (defined as the proportion of women who self-collect a sample). Acceptability of intervention materials and self-sampling procedures will be measured using self-report surveys at follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Hispanic/Latina ethnicity
* Assigned female sex at birth
* Age 30-65, consistent with guidelines for HPV DNA testing for cervical cancer screening
* Speak and read English or Spanish
* Computer or other device with internet connection
* Overdue for cervical cancer screening (e.g., no cytology-based screening within the past 3 years; no hrHPV testing either alone or in combination with cytology in the past 5 years).

Exclusion Criteria:

* Prior diagnosis of cervical cancer or abnormality (e.g., dysplasia)
* Had a hysterectomy/removal of the cervix
* Compromised immune system (e.g., known HIV)
* Women who self-report that they are pregnant or are within three months after a pregnancy

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Intervention Feasibility | 1 month
  The number of participants in the intervention arm who attend at least one session

SECONDARY OUTCOMES:
Participation in screening | 1 month
  The number of participants who return a self-collected sample

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Fang, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data and associated documentation can be made available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. All procedures will be compliant with NIH regulations on the distribution of unique research resources.

REFERENCES:
- [Derived] Fang CY, Cora-Cruz M, Koirala P, Perez S, Li M, Egleston BL, Chen Y, Mantia-Smaldone G, Martinez O. Juntas Contra el Virus del Papiloma Humano: protocol for a pilot randomized controlled trial of an HPV self-sampling intervention for underscreened Latinas. Pilot Feasibility Stud. 2025 May 10;11(1):65. doi: 10.1186/s40814-025-01648-y. PMID 40349085